CLINICAL TRIAL: NCT03383029
Title: Evaluation of the Feasibility and Preliminary Efficacy of the Parent-Mediated Integrated Eating Aversion Treatment (iEAT) Manual
Brief Title: iEAT 2.0 Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lindsey Burrell, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00099562
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Gastrointestinal Disorders
Keywords: Nutrition; Behavioral
MeSH Terms: conditions — Gastrointestinal Diseases; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iEAT (Experimental): Children with food refusal will participate in the iEAT program.
  Interventions: Behavioral: iEAT Program

INTERVENTIONS:
Behavioral: iEAT Program — The iEAT Program is a six-month long behavioral intervention consisting of 10 biweekly outpatient appointments of about 1 hour in length. The iEAT manual will guide behavioral intervention targeting severe feeding disorders and will involve some combination of escape extinction, reinforcement, and antecedent manipulation of food presentation to lessen the aversive quality of the meal.

SUMMARY:
The purpose of this study is to learn more about the eating behaviors of children with chronic food refusal. Specifically, investigator's aim to see how the integrated Eating Aversion Treatment (iEAT) may affect a child's food consumption. The manual is a structured multidisciplinary treatment, including a psychologist and dietitian with consultation from a speech-language pathologist. The treatment is designed to increase the volume of foods a child eats and decrease their reliance on a feeding tube or formula. The manual includes informational handouts, data collection forms, and instructions to guide the increase in feeding demands while reducing reliance on formula to meet a child's nutritional needs.

Children with chronic food refusal will participate in this study at the Marcus Autism Center. All children who enroll will receive the iEAT treatment. This involves 10 bi-weekly sessions that last approximately one hour, over the course of 5 months and a 1 month follow-up visit. Therefore, the study will last a total of 6 months.

DETAILED DESCRIPTION:
This study seeks to further the development of iEAT by including participants that demonstrated improvements in a previously conducted pilot study, and finalize the treatment manual to include the standardized decision rules to increase feeding demands, further integrate the multidisciplinary team (nutrition and speech pathology), and include supplementary sessions to better address individual treatment needs.

Investigators propose to enroll participants with chronic food refusal and formula or feeding tube dependence. Treatment will involve 10 biweekly outpatient appointments and 1 follow-up appointment of about 1 hour in length. Assessment and treatment will involve a multidisciplinary team including behavioral psychology, speech pathology and nutrition. Target behaviors including grams consumed, percent dependence on formula/feeding tube, and the clinical global impression scale, which will be assessed during a meal observation, 3-day food record, and evaluation with the dietitian and independent evaluator. Participants will be assessed pre-treatment, mid-treatment, and post-treatment and complete a one month follow-up to assess long term effects.

ELIGIBILITY:
Inclusion Criteria:

* Present with partial food refusal as evidenced by greater than 75% of caloric needs met by bottle, formula, or tube feedings
* Have a medical history significant for an organic factor (e.g., gastrointestinal issues) which influenced the development of feeding concern
* Safe to consume up to 100% of his/her needs orally
* Parents of subjects must be English literate
* Ability to complete at least 2 structured meals each day

Exclusion Criteria:

* Active medical diagnoses requiring hospitalization or significant oversight from a physician
* Active medical, structural, or functional limitations preventing safe oral intake of pureed foods

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Change in Percent Oral Intake | Baseline, Post-Intervention (Week 20)
  Oral intake will be assessed through the three-day food diary on which parents will record the child's daily intake. The percent of needs consumed orally will be reported.
Change in Total Oral Grams Consumed During Meal | Baseline, Post-Intervention (Week 20)
  Total oral grams consumed during a meal will be rated by trained observers captured by the meal observation form and collected during study visits.
Change in Percent Needs Met by Formula or Feeding Tube | Baseline, Post-Intervention (Week 20)
  Formula and feeding tube intake will be assessed through the three-day food diary on which parents will record the child's daily intake. The percent of needs consumed via bottle or tube will be reported.
Clinical Global Impression Scale - Improvement (CGI-I) Score | Post-Intervention (Week 20)
  The CGI-I is a seven-point scale measure of overall change from baseline. Scores will be ranked from 1 (Very Much Improved) through 4 (Unchanged) to 7 (Very Much Worse). Scores of "Much Improved" or "Very Much Improved" will be used to define positive responses; all other scores will indicate negative responses. Total scores range from 1 to 7; where 1 indicates the most improvement and 7 indicates greatest worsening.

SECONDARY OUTCOMES:
Change in Parenting Stress Index (PSI) Score | Baseline, Post-Intervention (Week 20)
  The PSI is a 36-item measure completed by a parent or caregiver designed to screen for stress in the parent-child relationship, identifying dysfunctional parenting and child adjustment problems. Raw scores are converted into percentile scores. A score which falls between the 15th and 80th percentile is considered typical. High scores are those at or above the 85th percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Burrell, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States